CLINICAL TRIAL: NCT00713557
Title: Phase 4 Study to Compare Different Therapeutic Strategies for Patients With ACS
Brief Title: Shanghai Registry of Acute Coronary Events
Status: Terminated | Type: Observational
Why Stopped: devices applied in the study were no more available in the market, and medical intervention section was completed.
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government); Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Qi, MD, MD, Shanghai Jiao Tong University School of Medicine
Other Study IDs: RJH
Record Dates: First submitted 2008-07-07; First posted 2008-07-11 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
Keywords: coronary angioplasty
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome | interventions — Drug-Eluting Stents; Tirofiban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- 1: patients with acute ST-elevation myocardial infarction and receiving primary percutaneous coronary intervention Subgroup: Patient Transferring vs. Physician Transferring strategy
  Interventions: Device: drug-eluting stent
- 2: patients with acute ST-elevation myocardial infarction treated by thrombolysis or facilitated PCI Subgroup: upstream use of Tirofiban + primary PCI vs. downstream use of tirofiban + primary PCI
  Interventions: Device: drug-eluting stent; Drug: Tirofiban
- 3: patients with non-ST-elevation ACS treated by immediate PCI
  Interventions: Device: drug-eluting stent
- 4: patients with non ST-elevation ACS treated by elective PCI
  Interventions: Device: drug-eluting stent
- 5: STEMI patient with multivessel disease, complete revascularization is planned to achieve during the index hospitalization.i.e.P-PCI for culprit lesion,combined with staged PCI for remaining diseased vessel.
- 6: STEMI patient with multivessel disease, complete revascularization is planned to achieve at 6 weeks after STEMI onset.i.e.P-PCI for culprit lesion during index hospitalization,combined with staged PCI for remaining diseased vessel at 6-week's follow-up(secondary hospitalization).

INTERVENTIONS:
Device: drug-eluting stent — drug-eluting stent, including sirolimus-eluting, paclitaxel-eluting and other types of China-made drug-eluting stent
  Other Names: Cypher stent; Taxus stent; Firebird stent; Excel stent
  Groups: 1; 2; 3; 4
Drug: Tirofiban — upstream (in emergency room) versus downstream (in catheterization lab) intra-coronary loading versus conventional intravenous loading
  Groups: 2

SUMMARY:
SRACE is an multicenter observational database of outcomes for patients who are hospitalized with an acute coronary events. SRACE includes over 20 hospitals in Shanghai China that have enrolled a total of more than 3,000 patients since 2005, with an annual enrollment of 500 patients. The major purpose of the SRACE program is to evaluate the prognosis of patients admitted to the hospital due to acute coronary events, comparing different therapeutic strategies, in-hospital transferring system, and so on. All participating physicians receive confidential quarterly reports showing ther outcomes side-by-side with the aggregate outcomes of all participating hospitals.

DETAILED DESCRIPTION:
consecutive patients with STEMI who presented symptoms within 12 hours and treated by primary PCI in Shanghai, were enrolled in the prospective sysytem. Several strategies were applied in these patients, including physician vs. patient transfer strategy, upsteam vs. downstream strategy, Firebird stent vs. Excel stent (bio-absorbable SES), etc. Once the patient was randomized to one of these study, he will be denied to the others. Clinical and angiographic outcomes were compared, with the final purpose to find an optimal strategy in treating AMI patients.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the hospital with acute coronary syndrome and received medical or interventional treatment

Exclusion Criteria:

* non ACS patients;
* complicated with other lethal disease
* predicted life span less than 12 months
* known allergy history to any anti-platelet or anti-thrombin medicine
* unconscious at the time of arrival at the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to the hospital with acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2005-03; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiac events(MACE), including death, non-fatal re-MI, and target vessel revascularization | in-hospital, 30d, and long-term follow-up

SECONDARY OUTCOMES:
stroke, stent thrombosis | in-hospital, 30d, and long-term follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Wei Feng Shen, MD,PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Dept. of Cardiology, Ruijin Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Zhang Q, Zhang RY, Qiu JP, Zhang JF, Wang XL, Jiang L, Liao ML, Zhang JS, Hu J, Yang ZK, Shen WF. Prospective multicenter randomized trial comparing physician versus patient transfer for primary percutaneous coronary intervention in acute ST-segment elevation myocardial infarction. Chin Med J (Engl). 2008 Mar 20;121(6):485-91. PMID 18364130
- [Result] Zhang Q, Zhang RY, Qiu JP, Zhang JF, Wang XL, Jiang L, Liao ML, Zhang JS, Hu J, Yang ZK, Shen WF. One-year clinical outcome of interventionalist- versus patient-transfer strategies for primary percutaneous coronary intervention in patients with acute ST-segment elevation myocardial infarction: results from the REVERSE-STEMI study. Circ Cardiovasc Qual Outcomes. 2011 May;4(3):355-62. doi: 10.1161/CIRCOUTCOMES.110.958785. Epub 2011 Apr 26. PMID 21521833
- [Result] Qiu JP, Zhang Q, Lu JD, Wang HR, Lin J, Ge ZR, Zhang RY, Shen WF. Direct ambulance transport to catheterization laboratory reduces door-to-balloon time in patients with acute ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention: the DIRECT-STEMI study. Chin Med J (Engl). 2011 Mar;124(6):805-10. PMID 21518584
- [Derived] Zhang Q, Qiu JP, Kirtane AJ, Zhu TQ, Zhang RY, Yang ZK, Hu J, Ding FH, DU R, Shen WF. Comparison of biodegradable polymer versus durable polymer sirolimus-eluting stenting in patients with acute st-elevation myocardial infarction undergoing primary percutaneous coronary intervention: results of the RESOLVE study. J Interv Cardiol. 2014 Apr;27(2):131-41. doi: 10.1111/joic.12102. PMID 24697948